CLINICAL TRIAL: NCT06110182
Title: Evaluation of the Advantage in the Use of Enteral Nutrition in Children Treated for Acute Lymphoblastic Leukemia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, DEUTSCH Hélène, Dr Hélène DEUTSCH, Central Hospital, Nancy, France
Other Study IDs: 2023_PI_069
Record Dates: First submitted 2023-10-26; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Leukemia, Lymphoblastic
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- enteral nutrition: children who received enteral nutritional support during treatment
  Interventions: Dietary Supplement: enteral or parenteral nutritional support
- parenteral nutrition: children who received parenteral nutritional support during treatment
  Interventions: Dietary Supplement: enteral or parenteral nutritional support

INTERVENTIONS:
Dietary Supplement: enteral or parenteral nutritional support — Parents will be classified based on whether they received enteral or parenteral nutritional support during treatment.

SUMMARY:
This is a multicenter retrospective study (Reims and Nancy), with data collection over 12 years from 01/01/2010 to 12/31/2022 Patients included are children diagnosed with acute lymphoblastic leukemia between 2010 and 2021 in the 2 centers.

Patients will be categorized into 3 groups:

* No nutritional support
* Support by enteral nutrition
* Parenteral nutrition support Their nutritional status will be assessed at the end of induction, at 6 months and then at 12 months from diagnosis.

The main objective of this study is therefore to compare the nutritional status of children with acute lymphoblastic leukemia depending on whether they received enteral or parenteral nutritional support during their treatment.

The secondary objective is to evaluate the occurrence of complications during treatment according to the nutritional support received.

ELIGIBILITY:
Inclusion Criteria:

* Children between 1 and 18 years old diagnosed with Medium risk/ High Risk B acute lymphoblastic leukemia or Standard/ High Risk T acute lymphoblastic leukemia between 2010 and 2021 in Nancy and Reims.

Exclusion Criteria:

* Patients less than 1 year old
* leukémia with philadelphia chromosome
* standard risk B acute lymphoblastic leukemia
* bone marrow transplant during treatment
* death during the year following diagnosis
* refusal of the patient (parents) to participate in the study

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children diagnosed with acute lymphoblastic leukemia between 2010 and 2021 in Nancy and Reims
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Z-score | 6 months
  Compare the improvement in Z-score between the date of diagnosis and 6 months from diagnosis in children using parenteral nutrition and those using enteral nutrition during treatment of their acute lymphoblastic leukemia

SECONDARY OUTCOMES:
BMI | 6 months
  Compare the improvement in BMI between the date of diagnosis and 6 months from diagnosis in children using parenteral nutrition and those using enteral nutrition during treatment of their acute lymphoblastic leukemia
albumin | 6 months
  Compare the improvement in albumin level between the date of diagnosis and 6 months from diagnosis in children using parenteral nutrition and those using enteral nutrition during treatment of their acute lymphoblastic leukemia
complications | 1 year
  Compare the percentages of occurrence of complications between the date of diagnosis and 6 months after diagnosis in children using parenteral nutrition and those using enteral nutrition during treatment for their acute lymphoblastic leukemia

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, France